CLINICAL TRIAL: NCT06065579
Title: Efficacy of Well-Being Promotion Program for Management of Emotional and Behavioural Among Adolescents
Brief Title: Efficacy of Well-Being Promotion Program for Management of Emotional and Behavioural Problems Among Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Madiha Arshad, Efficacy of Well-Being Promotion Program for Management of Emotional and Behavioural Problems Among Adolescents, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JinnahWU
Record Dates: First submitted 2023-09-23; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Well-being, Emotional and Behavioral Problems, Adolescents
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group will receive intervention
  Interventions: Other: Well-Being Promotion Program
- Control Group (No Intervention): Control group will not receive intervention

INTERVENTIONS:
Other: Well-Being Promotion Program — the well-being promotion program (Suldo,2016) , an intervention designed to improve subjective well-being. It was postulated that this intervention will eventually assist in managing emotional and behavioural problems among adolescents enrolled in the program.
  Arms: Intervention Group

SUMMARY:
The objectives of the study are given as under;

1. To examine the efficacy of the Well-being Promotion Program in enhancing subjective well-being, positive affect, life satisfaction and reducing emotional /behavioral problems , negative affect among adolescents with emotional and behavioral problems.
2. To examine the differences in terms of subjective well-being, emotional / behavioral problems , positive / negative affect and life satisfaction between the treatment and control group after intervention.
3. To examine the differences in terms of subjective well-being, emotional / behavioral problems, positive / negative affect and life satisfaction in the intervention group at (T1) before and at (T2) after intervention.

DETAILED DESCRIPTION:
In this study, adolescents within age range ( 14-19years) will participates in the study because this study focus on the emotional and behavioral problems and their low level of well-being and life satisfaction among adolescents. Adolescence is a developmental period in which dramatically emotional changes occur which may be the result of biological changes such as secretions of hormones. Chances of psychological distress are increased due to emotional changes. Depression and anxiety are most common psychopathology in adolescents (Ma & Fang, 2019). Child turns out to be independent, gradually deals with the external world and starts taking his/her decisions such as selection of subjects, peer pressure and so on. Thus , it is important to focus on mental health and management of emotional and behavioral problems.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria Only those participants who meet the category of moderate level of emotional and behavioural problems through Strength and difficulty Questionnaire (SDQ; Urdu Version) (Samad et al., 2005) will be selected for the study.

Exclusion Criteria:

* Exclusion Criteria Those participants who meet high levels of emotional and behavioural problems through Strength and difficulty Questionnaire (SDQ; Urdu Version) (Samad et al., 2005) will not be selected for the study.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Emotional and Behavioural Problems Among Adolescents | 2.5 months
  Emotional and behavioural problems will be measured through the Strength and Difficulty Questionnaire(SDQ- Urdu Version) (Samad et al., 2005). High score on the Strength and Difficulty Questionnaire(SDQ- Urdu Version indicates more emotional and behavioural Problems .

CONTACTS AND LOCATIONS:
Locations (1):
- Madiha Arshad, Sukkur, Pakistan

IPD SHARING:
Plan to Share IPD: No